CLINICAL TRIAL: NCT03801174
Title: Using Partners to Enhance Long-Term Weight Loss
Acronym: Partner2Lose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Duke University (Other); RTI International (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-1400; 1R01DK111491-01A1 (NIH); A539722 (Other: University of Wisconsin, Madison); SMPH/SURGERY (Other: University of Wisconsin, Madison); 2018-1400-CP028 (Other: Most recent IRB approved protocol)
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partner-assisted intervention (Experimental): Patients and partners will receive intervention
  Interventions: Behavioral: Partner-assisted intervention
- Patient-only intervention (Active Comparator): Patients will receive intervention
  Interventions: Behavioral: Patient-only intervention

INTERVENTIONS:
Behavioral: Partner-assisted intervention — All patients will receive group-based weight loss program for 6 months featuring a calorie-restricted diet and physical activity. Then, all patients will receive a weight loss maintenance intervention for 12 months that involves maintenance-specific content, transitions to individual telephone calls, and decreases frequency of contact. Partners will attend some patient group sessions and be informed of patients' goals and relapse plans. Intervention will be withdrawn for the last 6 months to examine sustainability of effects.
  Arms: Partner-assisted intervention
Behavioral: Patient-only intervention — All patients will receive group-based weight loss program for 6 months featuring a calorie-restricted diet and physical activity. Then, all patients will receive a weight loss maintenance intervention for 12 months that involves maintenance-specific content, transitions to individual telephone calls, and decreases frequency of contact. Intervention will be withdrawn for the last 6 months to examine sustainability of effects.
  Arms: Patient-only intervention

SUMMARY:
This study involves an evaluation of the role of domestic partner support in a comprehensive weight loss initiation and maintenance program.

DETAILED DESCRIPTION:
Couples will be randomized to a comprehensive weight program directed at patients alone or involving their partners. In months 1-6, all patients will receive group-based weight loss program. In months 7-18, all patients will receive a telephone-based weight loss maintenance intervention. In the partner-assisted arm only, partners will participate in the intervention, learning and practicing communication skills and support strategies. In months 19-24, intervention will be withdrawn to examine sustainability of effects.

Due to COVID-19, option of doing screening and outcome assessment visits and attending the group classes (including exercise) remotely via a video conference may be available. COVID-19 survey will be administered every 3 month starting at screening/enrollment visit.

ELIGIBILITY:
Inclusion Criteria (patients):

* Aged 18-74 years
* BMI 27-29.9 kg/m2 plus at least one obesity-related comorbidity or BMI >=30 kg/m2
* Cohabitating and at least daily contact with a spouse/domestic partner
* Access to reliable transportation
* Desire to lose weight
* Speak and read English
* Agree to attend visits per protocol
* Score of at least 4 out of 6 on Callahan cognitive screener
* Able to stand without assistance for weight measurements without assistance
* Possess individual email address
* Possess individual smart phone with data and texting plan
* Able to complete online screener without assistance
* Able to use a smartphone, tablet or computer with a video camera or webcam and microphone to download apps and to connect to a video conference call without assistance

Exclusion Criteria (patients):

* Currently or planning to become pregnant or breastfeeding in the study timeframe
* Weight loss ≥ 5 lb in the month prior to screening
* Currently enrolled, or enrolled in previous 3 months, in a clinical or research program focusing on lifestyle change that could affect weight
* Significant dementia, schizophrenia, psychosis, or drug or alcohol abuse
* Chronic or unstable illness that would limit ability to participate (e.g., recent hospitalization; unstable heart disease in the 6 months prior to screening, chronic kidney disease stage 4 or higher)
* Living a nursing home or receiving visits from a home health care agency
* Planning to relocate in the next 2.5 years
* Current use of prescription or over-the-counter weight loss medications
* History of bariatric surgery or planning to have bariatric surgery in the study timeframe
* Impaired hearing
* Currently receiving, or received in the past 6 months, treatment for cancer other than skin cancer
* Use of insulin, sulfonylureas, or meglinitides for diabetes
* High diuretic dose
* Exertional chest pain, dizziness, or lightheadedness
* Pain or other condition than prohibits mild-moderate exercise
* History of ascites requiring paracentesis

Inclusion criteria (partner):

* Aged 18 or older
* Willing to participate
* Access to reliable transportation
* Speak and read English
* Score of at least 4 out of 6 on Callahan cognitive screener
* Possess smart phone with data and texting plan (not shared with index patient)
* Possess email address (not shared with index patient)
* Able to complete online screener without assistance

Exclusion criteria (partner):

* BMI <18.5 kg/m2
* Significant dementia, schizophrenia, psychosis, or drug or alcohol abuse
* Residing in a nursing home or receiving home health care
* Impaired hearing
* Currently receiving, or received in the past 6 months, treatment for cancer other than skin cancer
* Chronic or unstable illness that would limit ability to participate (e.g., recent hospitalization; unstable heart disease in the 6 months prior to screening)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Voils, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voils CI, Shaw RJ, Gavin KL, Hetzel SJ, Lewis MA, Pabich S, Johnson HM, Elwert F, Mao L, Gray KE, Yuroff A, Garza K, Yancy WS Jr, Porter LS. Outcomes from Partner2Lose: a randomized controlled trial to evaluate 24-month weight loss in a partner-assisted intervention. BMC Public Health. 2024 Jul 20;24(1):1948. doi: 10.1186/s12889-024-19464-z. PMID 39033273
- [Derived] Voils C, Shaw R, Gavin K, Hetzel S, Lewis M, Pabich S, Johnson H, Elwert F, Mao L, Gray K, Yuroff A, Garza K, Yancy W, Porter L. Primary outcomes from Partner2Lose: A randomized controlled trial to evaluate partner involvement on long-term weight loss. Res Sq [Preprint]. 2024 Mar 11:rs.3.rs-4001003. doi: 10.21203/rs.3.rs-4001003/v1. PMID 38559225
- [Derived] Miller HN, Voils CI, Cronin KA, Jeanes E, Hawley J, Porter LS, Adler RR, Sharp W, Pabich S, Gavin KL, Lewis MA, Johnson HM, Yancy WS Jr, Gray KE, Shaw RJ. A Method to Deliver Automated and Tailored Intervention Content: 24-month Clinical Trial. JMIR Form Res. 2022 Sep 6;6(9):e38262. doi: 10.2196/38262. PMID 36066936
- [Derived] Voils CI, Shaw R, Adler R, Jeanes E, Lewis MA, Sharp W, Cronin KA, Hetzel S, Mao L, Johnson HM, Elwert F, Pabich S, Gavin KL, Yancy WS Jr, Porter LS. Protocol for Partner2Lose: A randomized controlled trial to evaluate partner involvement on long-term weight loss. Contemp Clin Trials. 2020 Sep;96:106092. doi: 10.1016/j.cct.2020.106092. Epub 2020 Aug 1. PMID 32750431
- See also: Partner2Lose website — http://www.partner2lose.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment numbers reflect only patients, not dyads, as this is how the study analysis was powered.
Pre-assignment Details: Enrollment numbers reflect only patients, not dyads. Partners were not assessed and therefore are not their own arm. Partners were not considered as enrolled, and are not included in the reported enrollment number. Partners did not have Baseline, pre-specified Primary and/or Secondary Outcome Measure, and Adverse Event data collected.
Groups:
- Partner-assisted Intervention: Patient: Patients and partners will receive intervention
  Partner-assisted intervention: All patients will receive group-based weight loss program for 6 months featuring a calorie-restricted diet and physical activity. Then, all patients will receive a weight loss maintenance intervention for 12 months that involves maintenance-specific content, transitions to individual telephone calls, and decreases frequency of contact. Partners will attend some patient group sessions and be informed of patients' goals and relapse plans. Intervention will be withdrawn for the last 6 months to examine sustainability of effects.
Period: Overall Study
Arm/Group | Partner-assisted Intervention: Patient | Patient-only Intervention
Started | 115 | 116
Completed | 63 | 80
Not Completed | 52 | 36
Not completed — Withdrawal by Subject | 14 | 15
Not completed — Death | 1 | 0
Not completed — Pregnancy | 2 | 2
Not completed — Lost to Follow-up | 19 | 10
Not completed — Other | 4 | 3
Not completed — Lack of Efficacy | 4 | 0
Not completed — Unwilling to complete activities | 5 | 6
Not completed — Moved out of area | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected on partners.
Groups:
- Total: Total of all reporting groups
Arm/Group | Partner-assisted Intervention: Patient | Patient-only Intervention | Total
Number analyzed (Participants) | 115 | 116 | 231
Age, Continuous [Mean (Standard Deviation); unit: years]
  Participant | 47.3 (11.31) | 47.24 (11.76) | 47.27 (11.51)
Sex/Gender, Customized [Number; unit: participants]
  Identify as Female | 76 | 79 | 155
  Identify as Male | 37 | 37 | 74
  Genderqueer | 1 | 0 | 1
  Multi-gender | 1 | 0 | 1
  Birth sex - Female | 78 | 79 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 108 | 112 | 220
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 6 | 6 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 97 | 101 | 198
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 115 | 116 | 231
Body weight [Mean (Standard Deviation); unit: kilograms] | 106.20 (19.03) | 106.90 (19.84) | 106.55 (19.41)
Daily caloric intake [Mean (Standard Deviation); unit: kcal/day] | 2182.66 (730.00) | 2103.10 (737.88) | 2142.88 (733.43)
Steps per day [Mean (Standard Deviation); unit: steps/day] | 8023.37 (3412.32) | 8203.70 (3622.56) | 8114.40 (3512.68)

OUTCOME MEASURES:

1. Primary Outcome: Body Weight (kg)
Description: Measured on a calibrated, digital scale to the nearest 0.1 kg, assessed every 6 months with 24 months as primary endpoint
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Partner-assisted Intervention | Patient-only Intervention
Number analyzed (Participants) | 115 | 116
kilograms | 104.46 [101.73 to 107.18] | 104.23 [101.54 to 106.92]
Statistical Analysis 1: Comparison: Partner-assisted Intervention vs Patient-only Intervention; Test type: Superiority; p = .804, Mixed Models Analysis; Mean Difference (Net) = -0.23, 95% CI 2-sided [-2.0 to 1.6], Standard Error of Mean 0.92

2. Secondary Outcome: Caloric Intake (kcal)
Description: average estimated daily intake from ASA24 Dietary Assessment Tool, assessed every 6 months with 24 months as primary endpoint
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: KCALs/day
Arm/Group | Partner-assisted Intervention | Patient-only Intervention
Number analyzed (Participants) | 115 | 116
KCALs/day | 1835 [1689 to 1980] | 1885 [1746 to 2024]
Statistical Analysis 1: Comparison: Partner-assisted Intervention vs Patient-only Intervention; Test type: Superiority; p = .590, Mixed Models Analysis; Mean Difference (Net) = 50.2, 95% CI 2-sided [-132 to 233], Standard Error of Mean 93.0

3. Secondary Outcome: Physical Activity
Description: average daily steps over past 7 days from Fitbit, assessed every 6 months with 24 months as primary endpoint
Time Frame: 24 months
Measure: Mean (95% Confidence Interval); unit: steps/day
Arm/Group | Partner-assisted Intervention | Patient-only Intervention
Number analyzed (Participants) | 115 | 116
steps/day | 7400 [6615 to 8186] | 8206 [7475 to 8936]
Statistical Analysis 1: Comparison: Partner-assisted Intervention vs Patient-only Intervention; Test type: Superiority; p = .069, Mixed Models Analysis; Mean Difference (Net) = 806, 95% CI 2-sided [-64 to 1675], Standard Error of Mean 443

4. Other Pre Specified Outcome: Transformation of Motivation for Diet
Description: Score based on 12-item Unidimensional Relationship Closeness Scale (1-7, strongly disagree to strongly agree) and single-item Inclusion of Other in Self scale (7 Venn diagrams)
Time Frame: 3 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Outcome Efficacy for Diet
Description: 5 items assessed on 11-point scale ranging from 0 (not at all effective) to 10 (very effective)
Time Frame: 3 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Couple Efficacy for Diet
Description: 5 items assessed on 11-point scale ranging from 0 (not at all confident) to 10 (very confident)
Time Frame: 3 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Social Support for Diet
Description: 9 items assessed on 5-point scale (never, rarely, sometimes, often, almost always)
Time Frame: 3 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Use of Communal Coping Strategies for Diet
Description: 5 items assessed on 5-point frequency scale (never, sometimes, frequently, often, very often)
Time Frame: 3 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Transformation of Motivation for Physical Activity
Description: as for outcome 4
Time Frame: 3 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Outcome Efficacy for Physical Activity
Description: 5 items assessed on 11-point scale ranging from 0 (not at all effective) to 10 (very effective)
Time Frame: 3 months
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Couple Efficacy for Physical Activity
Description: 5 items assessed on 11-point scale ranging from 0 (not at all confident) to 10 (very confident)
Time Frame: 3 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Social Support for Physical Activity
Description: 9 items assessed on 5-point scale (never, rarely, sometimes, often, almost always)
Time Frame: 3 months
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Use of Communal Coping Strategies for Physical Activity
Description: 5 items assessed on 5-point frequency scale (never, sometimes, frequently, often, very often)
Time Frame: 3 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 24 months
Description: Partners were not assessed for adverse events.
Arm/Group | Partner-assisted Intervention | Patient-only Intervention
All-Cause Mortality (participants affected / at risk) | 1/115 | 0/116
Serious Adverse Events (participants affected / at risk) | 3/115 | 3/116
Other Adverse Events (participants affected / at risk) | 55/115 | 52/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partner-assisted Intervention (N=115) | Patient-only Intervention (N=116)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ablation (Cardiac disorders) | 0 (0) | 1 (1)
Death (Cardiac disorders) | 1 (1) | 0 (0)
Ulcerative colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse medication interaction (General disorders) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Hip replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Partner-assisted Intervention (N=115) | Patient-only Intervention (N=116)
Anemic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrinologist prescribed diet change (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Nonclassical congenital adrenal hyperplasia (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Burning mouth syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pravovirus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach ache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Ulcerative colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Common cold (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever and chills (General disorders) | 0 (0) | 1 (1)
Mouth pain (General disorders) | 1 (1) | 0 (0)
Swollen feet (General disorders) | 0 (0) | 1 (1)
Liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Bell's palsy (Infections and infestations) | 1 (1) | 0 (0)
Blood infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Common cold (Infections and infestations) | 7 (8) | 8 (12)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Flu (Infections and infestations) | 2 (3) | 7 (8)
Food poisoning (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Leg infection (Infections and infestations) | 0 (0) | 1 (1)
Post-surgical infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory infection (Infections and infestations) | 2 (2) | 1 (2)
Sinus infection (Infections and infestations) | 1 (1) | 2 (2)
Strep throat (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0)
Vomiting (Infections and infestations) | 0 (0) | 1 (1)
Broken ankle (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Broken arm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Broken ribs (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foot injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypercholesterolemia (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Investigations) | 0 (0) | 1 (1)
Gluten intolerant (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pre-diabetes diagnosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type II diabetes diagnosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ACL tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Frozen shoulder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heel spurs (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Knee arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee injury (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder calcium deposits (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder fibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Shoulder injury (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Sprained ankle (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Torn hamstring (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torn labrum (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cyst removed (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizzy spells (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Leg nerve pain (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Binge eating disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Depression and anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Depression medication change (Psychiatric disorders) | 1 (1) | 0 (0)
Obsessive compulsive disorder diagnosis (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep issues (Psychiatric disorders) | 1 (1) | 2 (2)
Bladder cancer (Renal and urinary disorders) | 1 (1) | 0 (0)
Kidney stone (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract burning (Renal and urinary disorders) | 0 (0) | 1 (1)
Amenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PCOS diagnosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostate surgery (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Covid-19 (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 4 (4)
Heavy breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Long Covid-19 symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Poison ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Tick bite (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Appendix removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Back surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Breast biopsy (Surgical and medical procedures) | 0 (0) | 1 (1)
Cataract surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Dental crown procedure (Surgical and medical procedures) | 0 (0) | 1 (1)
Gall bladder removal (Surgical and medical procedures) | 0 (0) | 2 (2)
Knee replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Knee surgery (Surgical and medical procedures) | 0 (0) | 2 (2)
Meniscus tear (Surgical and medical procedures) | 0 (0) | 1 (1)
Root canal (Surgical and medical procedures) | 1 (1) | 0 (0)
Toe surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)
Varicose vein surgery (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03801174/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/74/NCT03801174/ICF_000.pdf